CLINICAL TRIAL: NCT04657627
Title: FOODS: Food shOppers' sOcial meDia Study
Acronym: FOODS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Dr Oonagh Markey (Unknown); Alexandra Todd (Unknown)
Responsible Party: Principal Investigator, Amanda Daley, Professor Amanda Daley, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1544
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Eating Behaviour of Discretionary Foods; Cognitive Restraint of Eating; Physical Activity; Body Weight
Keywords: Nutrition labelling; Physical activity; Social media
MeSH Terms: conditions — Motor Activity; Body Weight

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of two groups for 13 weeks: (i) PACE plus calorie information intervention group or (ii) calorie-only information comparator group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACE plus calorie information intervention group (Experimental): PACE plus calorie information intervention group will receive PACE plus calorie information of discretionary foods via social media posts.
  Interventions: Behavioral: PACE plus calorie labelling information
- Calorie-only information comparator group (Active Comparator): Calorie-only information comparator group will receive calorie-only information of discretionary foods via social media posts.
  Interventions: Behavioral: Calorie-only labelling information

INTERVENTIONS:
Behavioral: PACE plus calorie labelling information — The intervention group will be exposed to PACE plus calorie labelling information via Instagram and Twitter social media posts every day for 13 weeks.
  Arms: PACE plus calorie information intervention group
Behavioral: Calorie-only labelling information — The comparator group will be exposed to calorie-only labelling information via Instagram and Twitter social media posts every day for 13 weeks.
  Arms: Calorie-only information comparator group

SUMMARY:
This study aims to assess the effects of a new approach to food labelling called physical activity calorie equivalent (PACE) labelling. PACE food labelling provides the public with information about how many minutes (or miles/kilometres) of physical activity (e.g. walking or running) are equivalent to the calories contained in foods.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* BMI of ≥ 18.5 kg/m2.
* ≤ 3kg weight loss in previous 6 months.
* Access and ability to use personal Twitter and/or Instagram account via own smartphone, computer or tablet device.
* Access to the internet.
* Access to a set of weighing scales.

Exclusion Criteria:

* Unable to read and understand English.
* Experienced in the last 12 months or currently undergoing any of the following conditions or illnesses: coronary heart disease (CHD), hypertension, heart failure, stroke/transient ischaemic attack, atrial fibrillation, type 2 diabetes, chronic obstructive pulmonary disease (COPD), painful condition, dementia and cancer.
* Had bariatric surgery.
* Pregnant, lactating or planning to become pregnant in the next 12 months.
* Parallel participation in another weight, dietary or physical activity intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Change in eating behaviour of discretionary foods at 13 weeks | Pre-baseline (one time point prior to randomisation) and post-intervention (one time point after week 13)
  Eating behaviour of discretionary foods will be assessed by a modified version of Online Food Frequency Questionnaire (eNutri FFQ), designed to measure habitual food intake. Participants will record frequencies of discretionary food and drink items eaten during the last month (e.g. "1/week" or "1/day").

SECONDARY OUTCOMES:
Cognitive restraint of eating | Pre-baseline (one time point prior to randomisation) and post-intervention (one time point after week 13)
  A modified version (R18) of the Three-Factor Eating Questionnaire (TFEQ) will be used to measure cognitive restraint.
Physical activity | Pre-baseline (one time point prior to randomisation) and post-intervention (one time point after week 13)
  Self-reported physical activity behaviour will be assessed using the 7-day International Physical Activity Questionnaire (IPAQ)
Body weight | Pre-baseline (one time point prior to randomisation), mid-intervention (week 7) and post-intervention (one time point after week 13)
  Weight will be self-reported via participants own weighing scales. Participants will electronically send via email photograph evidence of readings of their fasted morning weight from weighing scales, following standardised instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Daley, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No